CLINICAL TRIAL: NCT06435195
Title: Clinical Characteristics and Analysis of Pituitary Complex and Rare Diseases
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K5112
Record Dates: First submitted 2024-05-17; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Pituitary Diseases
MeSH Terms: conditions — Pituitary Diseases | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pituitary Complex and Rare Diseases: The Pituitary Complex and Rare Diseases cohort consists of patients diagnosed with various pituitary disorders, including but not limited to pituitary adenomas, craniopharyngiomas, Rathke's cleft cysts, sellar region germ cell tumors, cavernous sinus syndrome, and other diseases. Patients requiring surgical resection or biopsy of pituitary pathologies will undergo transsphenoidal surgery or craniotomy.
  Interventions: Procedure: Surgical Removal; Procedure: Biopsy

INTERVENTIONS:
Procedure: Surgical Removal — Resection of pituitary pathologies.
Procedure: Biopsy — Taking a small tissue or liquid sample from the pituitary pathologies and the affected area for examination and diagnosis

SUMMARY:
The goal of this observational study is to systematically describe the clinical characteristics and outcomes of patients with pituitary complex and rare diseases at Peking Union Medical College Hospital. The main questions it aims to answer are:

* What are the influencing factors and rates of remission?
* What are the comorbidities associated with these diseases?
* What are the perioperative events, radiological findings, and pathological features?

Researchers will compare different patient groups to see if there are significant differences in these outcomes.

Participants will:

* Undergo detailed clinical evaluations.
* Provide medical history and data for analysis.
* Participate in follow-up assessments to monitor disease progression and treatment outcomes.

DETAILED DESCRIPTION:
The study aims to provide a comprehensive analysis of pituitary complex and rare diseases at Peking Union Medical College Hospital. By leveraging a large cohort, the research will explore various clinical characteristics and outcomes. Specifically, the study will examine influencing factors and rates of remission, the presence of comorbidities, and perioperative events. Additionally, it will evaluate radiological findings and pathological features to better understand these conditions. Through this detailed investigation, the study seeks to enhance knowledge and inform clinical practice regarding the management and prognosis of pituitary complex and rare diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rare sellar diseases including but not limited to pituitary adenomas (such as Thyrotropin-secreting pituitary adenomas, GH-secreting adenomas), craniopharyngiomas, Rathke's cleft cysts, sellar region germ cell tumors, cavernous sinus syndrome, and other diseases
* Detailed medical history, including clinical symptoms, treatment plans and follow-up outcomes

Exclusion Criteria:

* Incomplete medical records, especially missing key imaging diagnostic results
* Patients with coexisting primary central nervous system diseases unrelated to sellar region diseases (such as severe traumatic brain injury)
* Patients whose sellar region pathological diagnosis was changed or overturned during the follow-up period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are diagnosed with Pituitary Complex and Rare Diseases at Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Remission | Postoperative one week and extends to the latest follow-up, estimated at up to 3 years
  Hormonal normalization and free of pathologies

SECONDARY OUTCOMES:
Disease Comorbidities | From patient admission to an evaluation period extending up to the latest follow-up, estimately up to 3 years
  Systemic changes accompanied with Pituitary Complex and Rare Diseases
Postoperative complications | Postoperative one week and extends to the latest follow-up, estimated at up to 3 years
  adverse events or medical issues that arise after a surgical procedure on the pituitary diseases.These complications can include various problems such as bleeding, infection, hormonal imbalances, cerebrospinal fluid leaks, vision changes, or neurological deficits

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yao, MD, Principal Investigator — Department of Neurosurgery, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China